CLINICAL TRIAL: NCT05629195
Title: Study on the Influence of Skin Laxity on the Application Effect of Different PICC Catheterization Methods
Brief Title: The Effect of Skin Laxity on the PICC
Acronym: PICC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Yingshan Zheng, nurse, First People's Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: foshan202271
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Complications; Catheter

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tunneled PICC (Experimental): Placement of PICC catheter through tunnel technology
  Interventions: Device: tunneled PICC
- conventional PICC (Active Comparator): Placement of PICC catheter through conventional technology
  Interventions: Device: tunneled PICC

INTERVENTIONS:
Device: tunneled PICC — PICC catheter is inserted into the superior vena cava through the upper brachial vein by establishing a subcutaneous tunnel

SUMMARY:
To evaluate the clinical effect of tunneled PICC by comparing the rate of complications of the two groups of patients (tunneled PICC vs conventional PICC).

DETAILED DESCRIPTION:
In this study, tunneled PICC was compared with conventional PICC. Eligible subjects were randomly enrolled into the test group or control group by randomization (1:1), and observed and evaluated the occurrence of complications during and 7 ± 3 days, 30 ± 7 days, 60 ± 10 days, 90 ± 10 days, 120 ± 10 days (if any) after surgery and extubation at the end of treatment. To evaluate the clinical effect of tunneled PICC by comparing the rate of complications of the two groups of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old;
* Patients who need PICC catheterization according to the doctor's advice;
* There is no history of venous thrombosis, compression or blockage of superior vena cava, severe coagulation dysfunction and other contraindications for PICC catheterization;
* There is no serious cardiovascular disease, such as atrial fibrillation, pulmonary heart disease and other patients with abnormal P wave, and severe heart block before catheterization
* Patients who have not participated in other clinical studies;
* Patients who voluntarily participate in this clinical study and can cooperate with clinical follow-up

Exclusion Criteria:

* Known allergy to catheter material;
* The puncture site has a history of infection, injury and radiotherapy;
* The puncture site has a history of venous thrombosis or surgery;
* Severe abnormal bleeding and coagulation function;
* Superior vena cava compression syndrome;
* Surgical side limbs of breast cancer patients undergoing radical mastectomy or axillary lymph node dissection;
* The ipsilateral limb of the pacemaker and the arteriovenous fistula;
* patient or her/his family members refuse to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
rate of PICC complications | 120 days
  Including bleeding, subcutaneous congestion, lymphatic exudation, phlebitis (mechanical phlebitis, thrombophlebitis), infection (local infection, tunnel infection, catheter related blood flow infection), thrombus (symptomatic thrombus, asymptomatic thrombus), catheter ectopic, medical adhesive related skin damage, catheter damage and blockage, etc

SECONDARY OUTCOMES:
time of PICC insertion | 1 hour
  Time from the start of skin disinfection to the end of dressing fixation
Success rate of catheterization | 1 hour
  Judgment of successful catheterization: The catheterization is successful and the catheter is placed in an accurate position, that is, the tip of the catheter reaches within 1/3 of the lower part of the superior vena cava or near the junction of the right atrium.
score of operation pain | 1 hour
  Wong Banker facial expression scale was used. This method uses 6 facial expressions from smile to cry to express the degree of pain: 0 points for no pain, 1 point for slight pain, 2 points for some pain, 3 points for very pain, 4 points for severe pain, and 5 points for unbearable pain
rate of unplanned extubation | 120 days
  Extubation after abnormal treatment
rate of difficulty in decannulation | 120 days
  Probability of failure to pull out PICC due to vasospasm, adhesion with thrombus, wrapping of fibrin sheath, etc